CLINICAL TRIAL: NCT02759679
Title: Canine-Assisted Profiling of Lung Cancer From Human Breath
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: REK_2013/2053
Record Dates: First submitted 2016-03-17; First posted 2016-05-03 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung cancer (Other): Patients with lung cancer
  Interventions: Other: Human breath samples
- Controls (Other): Controls being either healthy or having other lung disease
  Interventions: Other: Human breath samples

INTERVENTIONS:
Other: Human breath samples

SUMMARY:
The study aims to optimize and define a reproducible and non-invasive method for canine assisted lung cancer detection, using human breath samples from patients and controls for training and testing purposes.

ELIGIBILITY:
Inclusion criteria:

Healthy volunteers, lung cancer or other lung disease.

Exclusion criteria:

Other known malignancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for lung cancer, of canines sniffing breath samples | 2 years
  Patients and Controls deliver breath samples to be presented for dogs in a Remote facility. Outcomes will be reported for individual dogs and combinations of dogs.

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Fløtten, MD, Principal Investigator — Haukeland University Hospital, Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No